CLINICAL TRIAL: NCT01831908
Title: The "Know Your Numbers" Program in Atahualpa - An Interventional Study Aimed to Reduce Cardiovascular Diseases and Stroke Burden in Rural Coastal Ecuador.
Brief Title: The "Know Your Numbers" Program in Atahualpa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clínica Kennedy (Other)
Collaborators: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Oscar H. Del Brutto, MD, Principal Investigator, The Atahualpa Project, Hospital Clínica Kennedy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAP-2013-03
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Risk Factors; Stroke; Ischemic Heart Disease
Keywords: cardiovascular health, stroke, ischemic heart disease
MeSH Terms: conditions — Stroke; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Sham Comparator): These persons will be advised on their cardiovascular status and will receive information on how to improve it.
  Interventions: Other: Lifestyle counseling
- People not seeking attention (No Intervention): Evaluation of cardiovascular health status will be performed in these persons as part of yearly door-to-door survey that will perform in Atahualpa up to the end of the study

INTERVENTIONS:
Other: Lifestyle counseling — People attending the community center will be provided with information on their health problems and will receive advise on how to improve blood pressure, glucose and cholesterol levels.
  Arms: Lifestyle counseling

SUMMARY:
Persons voluntarily attending the Community Center of the Atahualpa Project during one calendar year will be evaluated by trained personnel to check their cardiovascular health status. A chart with information of healthy behaviors as well as the numbers of the person's blood pressure, fasting glucose, and total cholesterol levels will be given. Persons who sign the informed consent will be visited at their homes after 3 months and than every year up to five years. The idea is to check whether the person followed our advises and if that compliance iis associated with improvement in the cardiovascular status or with a decreased incidence of stroke and ischemic heart disease, when compared with persons who did not attend the community center or those who did not follow our advices.

DETAILED DESCRIPTION:
Campaigns aimed to increase the level of awareness on cardiovascular risk factors may encourage people to change their lifestyles and to increase compliance with medication. This intervention has been called the "know your numbers program" and has been tested in developed countries. No study have evaluated the efficacy of this program in reducing the prevalence of ischemic heart disease and stroke on the long-term follow-up, and this program has not been applied to people living in rural areas of developing countries. During the study years, a community center of the Atahualpa Project will be open and stuffed with trained paramedical personnel that will attend people that voluntarily look for information. All these persons will be invited to participate in the "know your numbers" program, and those who sign the informed consent form will be enrolled in the program. Recruitment will be during one calendar year to assure the inclusion of a significant sample size of the population. As part of the initial visit, the CVH status of all individuals will be evaluated. Thereafter, persons will be informed on their health status and the best ways to improve it according to specific situations. Those who merit treatment for a given condition will be instructed to go to the physician for proper advice and prescription. A chart containing information on stroke and ischemic heart disease warning signs, as well as on healthy behaviors will be provided to all persons. All enrolled persons will be visited at their homes three months after the initial visit to the community center, and then, every year up to five years. We will evaluate whether the person followed our advices or the reasons for poor compliance. Persons will be asked to tell us if they remember the ischemic heart disease and stroke warning signs. Anthropometric parameters, blood pressure, total cholesterol and fasting glucose levels will be recorder at every visit and, again, any specific advice to improve "their numbers" or to seek for medical attention will be given. By the end of the study, the investigators will be able to correlate the CVH status of the person as well as the occurrence of vascular outcomes or death according to whether our advices were followed or not. Statistical analysis will be directed to refute the null hypothesis that this intervention does not improve the CVH and does not reduce the risk of stroke or ischemic heart disease

ELIGIBILITY:
Inclusion Criteria:

* Atahualpa residents aged 40 years or more who seek for information at the Atahualpa Community Center and sign the informed consent.

Exclusion Criteria:

* People not attending the Community Center or not signing the informed consent.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Improvement in cardiovascular health | 5 year

SECONDARY OUTCOMES:
Reduction in incident cases of stroke | 5 years

OTHER OUTCOMES:
reduction in incident cases of ischemic heart disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar H Del Brutto, MD, Principal Investigator — Universidad Espiritu Santo
Locations (1):
- Community Center, Atahualpa, Santa Elena, Ecuador

REFERENCES:
- [Background] Del Brutto OH, Penaherrera E, Ochoa E, Santamaria M, Zambrano M, Del Brutto VJ; Atahualpa Project Investigators. Door-to-door survey of cardiovascular health, stroke, and ischemic heart disease in rural coastal Ecuador--the Atahualpa Project: methodology and operational definitions. Int J Stroke. 2014 Apr;9(3):367-71. doi: 10.1111/ijs.12030. Epub 2013 Mar 19. PMID 23506643
- [Background] Del Brutto OH, Dong C, Rundek T, Elkind MS, Del Brutto VJ, Sacco RL. Cardiovascular health status among Caribbean Hispanics living in Northern Manhattan and Ecuadorian natives/mestizos in rural coastal Ecuador: a comparative study. J Community Health. 2013 Aug;38(4):634-41. doi: 10.1007/s10900-013-9658-0. PMID 23456686
- [Background] Del Brutto OH, Santamaria M, Ochoa E, Penaherrera E, Santibanez R, Pow-Chon-Long F, Zambrano M, Del Brutto VJ. Population-based study of cardiovascular health in Atahualpa, a rural village of coastal Ecuador. Int J Cardiol. 2013 Sep 30;168(2):1618-20. doi: 10.1016/j.ijcard.2013.01.017. Epub 2013 Feb 11. No abstract available. PMID 23410492